CLINICAL TRIAL: NCT04401930
Title: Eating Habits and Lifestyle Profile of an Italian Aging Cohort
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Hellas Cena, Tenured researcher, University of Pavia
Other Study IDs: 13052020; CUP E47F17000020009 (Other Grant/Funding Number: Regione Lombardia - POR FESR 2014-2020)
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Aging; Healthy Aging; Life Style; Eating Habit; Nutritional Deficiency; Sarcopenia
Keywords: elderly; life style; eating habits; health status; body composition; sarcopenia; nutritional deficiency; aged
MeSH Terms: conditions — Feeding Behavior; Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Free-living elderly: Free-living elderly over the age of 65 living in Metropolitan Area of Milan, in apparent good health conditions.
  Male and Female

SUMMARY:
Aging is characterized by low-grade inflammatory state, supported by impairment oxidative balance and endocrine changes, leading to changes in: body composition, such as decrease in lean body mass and increase in adipose tissue; resting metabolic rate; immune function; cognitive impairment. According to the Academy of Nutrition and Dietetics all subjects over the age of 60 should be able to access to adequate nutrition and appropriate nutritional services.

In order to ensure healthy aging and to reduce effects of specific diseases, recommendations are needed for illness and disability in this population, as well as adequate physical activity and specific support programs, culturally accepted.

The aim of this study is to evaluate eating habits in term of food consumption, health state and lifestyle in a sample of free-living elderly over the age of 65, living in Milan and surroundings.

In particular, profiling of the elderly population is performed using a survey in which information are collected on methods, contexts, time and ability to buy, prepare, consume and dispose of and recycle food. Eating habits and knowledge about food are detected through the analysis of food consumption frequencies, and lifestyle by assessing the level of physical activity, quality of sleep, smoking habit. Weight status and health status are evaluated through anthropometric measurements, body composition (bioelectrical impedance) and strength test.

Other information relating to social participation and other socio-demographic variables (age, gender, family composition, socio-economic status) are collected to have a completed profiling of target population.

Achieved results will help us to identify factors on which acting to ensure healthy aging and counteract inflammaging, the chronic low-grade systemic inflammation characteristic in the aging process.

Moreover, the study allows increasing the knowledge related to the needs and requirements of the target population to determine a good food policy and to increase the elderly empowerment.

DETAILED DESCRIPTION:
The study concerns the elderly population of the Milan Metropolitan Area. The aim is to identify and interpret the nutritional needs of the target population and thus implement the quality of life and the nutritional status of citizens through the evaluation of the dietary habits, health status and lifestyle of the elderly free-living.

The information is collected through a questionnaire consisting of 6 sections and includes batteries of questions and scales already validated in the literature: i) access to the points of sale; ii) consumer behavior; iii) eating habits; iv) opinions regarding accessibility; v) state of health, physical activity and sleep quality; vi) other socio-demographic information. The collected data will allow to identify different profiles of elderly people with respect to the investigated dimensions and to estimate the influence of different factors on eating habits and health status.

To complete the information collected with the questionnaire, functional and anthropmetric parameters are detected which are useful to complete the nutritional assessment of the target population. Specifically, the muscle strength, body composition, body weight, height, body circumferences, plicometry are measured, and the antripometric indices waist-height circumference ratio, waist-hip circumference ratio and arm muscle area are calculated.

SAMPLE SIZE: Based on the data on the population residing on 1 January 2017 from an Istat source, the residents of the metropolitan city of Milan aged 65 and over are 722703. The sample size was defined with the choice of a confidence level of 95% and of a confidence interval of 4%.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 65
* free-living
* autonomous, self sufficient
* acceptance and sign of informed consent

Exclusion Criteria:

* Age: under 65
* living in: nursing home, Extended Care
* hospitalized
* non autonomous, non self sufficient
* without acceptance and sign of informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Free-living over 65 subjects living in Milan and surroundings, in apparent good health conditions and self sufficient, able to express their consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the socio-demographic characteristics | 1 day
  Age, Educational level, family status, food safety, food security.
Assessment of eating habits | 1 day
  Eating habits: evaluated with the Food Habit (FHQ) section of questionnaire by Turconi et al. (2003), to investigate the eating habits related to daily number of meals, consumption of the main food groups (fruit, vegetables, etc) and soft drinks or alcoholic beverages. Each question has the following response: always, often, sometimes, never. The score assigned to each response ranged from 0 to 3, with the maximum score assigned to the healthiest one and the minimum score to the least healthy one according to the Italian National Dietary Guidelines (2018).
Assessment of smoking habits | 1 day
  Smoking habits: evaluated with specific semi-quantitative questions such as: "Are you smoker, no-smoker or former smoker?"; "How long have you been smoking?", "How old were you when you started smoking?" and "How many cigarettes do you smoke daily?" in current smokers; "How many years have passed since the last cigarette?" and "How many cigarettes per day did you use to smoke?" in former smokers. The minimum score was assigned to the healthiest habit.
Assessment of Physical activity level | 1 day
  Physical activity level evaluated with the International Physical Activity Questionnaires (IPAQ) - Short Form. The specific activity levels assessed are walking, moderate-intensity activities and vigorous-intensity activities. The scores are expressed in Metabolic Equivalent of task -minutes/week.The total score includes the sum of the duration (in minutes) and the frequency (days) of the three dimensions analyzed (walking, activity of moderate intensity and vigorous intensity). Higher number of MET per week relate with higher level of physical activity.
Assessment of Sleep Quality | 1 day
  Sleep Quality: evaluated with the Italian version of Pittsburgh Sleep Quality Index (PSQI), validated by Curcio et al (2011). It's a 19-item questionnaire investigating seven domains of sleep (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction). A global score, calculated from the score of each domains, higher than 5 is considered as an indicator of bad sleep quality.
Nutritional assessment: weight status | 1 day
  Measurement of: body weight in kilograms; height in centimeters, evaluated with prediction formula height-knee by Donini et al (2000); weight and height will be combined to report BMI in kg/m^2 to evaluate the weight status (underweight, normal, overweight, obesity);
Nutritional assessment: fat distribution | 1 day
  Measurement of: waist circumference in centimeters; hip circumference in centimeters; waist and hip will be combined to report waist-hip ratio (WHR) and waist and height will be combined to report waist-height ratio (WHtR), both as indicators of fat distribution and metabolic diseases risk.
Nutritional assessment: other antropometric parameters | 1 day
  Measurement of calf circumference in centimeters, as inidcator of muscle mass. Measurement of neck circumference in centimeters, as indicator of fat distribution and metabolic diseases risk.
Nutritional assessment: arm circumference and triceps skinfold thickness | 1 day
  Mesurement of: arm circumference in centimeters, as inidcator of muscle mass; triceps skinfold thickness in millimeters, as indicator of fatty mass; upper arm circumference and triceps fold will be combined to report the upper arm area in millimeters^2, upper arm muscle area in millimeters^2, upper arm fat area in millimeters^2.
Nutritional assessment: muscle strenght | 1 day
  Measurement of hand-grip in kilograms, to assess muscle strength
Nutritional assessment: body composition | 1 day
  Assessment of body composition with bioelectrical impedance analysis (BIVA).

SECONDARY OUTCOMES:
Adherence to Italian National Dietary Guidelines | 1 day
  Assess adherence to adequate eating habits from the analysis of Food Habits questionnaire according to the Italian National Dietary Guidelines.
Identify possible nutritional deficiencies | 1 day
  Identify possible nutritional deficiencies from the analysis of the Food Habits questionnaire
Lifestyle and nutritional status | 1 day
  Influence of eating habits analyzed with FHQ, sleep quality analyzed with PSQI, and physical activity level analyzed with IPAQ on nutritional status (all antropometric and body composition parameters collected).

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Lombardy, Italy